CLINICAL TRIAL: NCT05350709
Title: Comparison of the Effectiveness of Action Observation Therapy and Mirror Therapy on Upper Extremity Functions and Quality of Life in Patients With Parkinson's Disease.
Brief Title: Action Observation Therapy and Mirror Therapy in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Fatmanur Aybala KOÇAK, Medical Doctor, Physical Medicine and Rehabilitation Specialist, Principal Investigator, Associate Professor, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-02/02
Record Dates: First submitted 2022-04-18; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Parkinson Disease; Tremor
Keywords: mirror therapy; action observation therapy
MeSH Terms: conditions — Parkinson Disease; Tremor | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Investigator
Masking Description: via closed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mirror therapy (Active Comparator): An exercise program has been prepared for patients for use in mirror therapy. In this exercise program, firstly, joint movements of the hand and fingers (opening and closing the fingers one by one, making a fist, moving the hand to the right and left, turning the wrist) are shown. Then, activities with some small objects used in daily life (squeezing ball, putting clothespins, collecting paper clips from the table, using tongs, turning cards, turning pages) is shown. The patient will repeat the movement for 3 minutes. The patient will hold the affected extremity behind the mirror with the healthy extremity, the patient will look towards the affected side from the mirror and try to do the movements with the affected extremity. . The treatment period will be 20 sessions, 5 days a week, for 4 weeks.The exercises will take 1 hour, including half an hour of mirror therapy and half an hour of conventional exercises.
  Interventions: Other: mirror therapy
- action observational therapy (Active Comparator): An exercise video has been prepared for the patients to watch for the action observation therapy. In this video, first of all, joint movements of the hand and fingers (opening and closing the fingers one by one, making a fist, moving the hand to the right and left, turning the wrist, etc.) are shown. Then, activities with some small objects used in daily life (squeezing ball, putting clothespins, collecting paper clips from the table, using tongs, turning cards, turning pages, etc.). is shown. The patient will first watch the video of each movement, and then repeat the movement for 3 minutes. The treatment period will be 5 days a week, a total of 20 sessions for 4 weeks.The exercises will take 1 hour, including half an hour of action observational therapy and half an hour of conventional exercises.
  Interventions: Other: mirror therapy
- conventional therapy (Active Comparator): Conventional therapy includes range of motion exercises, walking and balance exercises. The treatment period will be 5 days a week, a total of 20 sessions for 4 weeks. The exercises will last for half an hour daily.
  Interventions: Other: mirror therapy

INTERVENTIONS:
Other: mirror therapy — 15 patients will be recruited to each group. Patients will receive a total of 20 sessions of treatment, 5 days a week.
  Other Names: action observational therapy; conventional therapy

SUMMARY:
Small muscles of the hand are affected due to involuntary movements and slowing of voluntary movements seen in Parkinson's disease. There is a loss of fine dexterity and coordination in the hand. It becomes difficult for patients to grasp and release of the objects. They become unable to perform daily activities such as buttoning up, holding keys, brushing teeth, holding forks, spoons and glasses, and writing. Therefore, a certain part of the rehabilitation program should be devoted to upper extremity rehabilitation. The aim of this study was to compare the effects of action observation therapy and mirror therapy, which have been used in the literature for many years, on upper extremity functions and quality of life in individuals with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older,
2. Diagnosed with idiopathic Parkinson's disease,
3. Parkinson's disease stage (patients with Hoehn Yahr≤3)
4. Patients who can hear and follow verbal instructions.

Exclusion Criteria:

1. Patients who cannot cooperate,
2. Patients with dementia or comorbidities affecting cognitive functions,
3. Patients with serious comorbidities (such as decompensated heart failure, decompensated kidney failure) and significant disability (such as vision loss, hearing loss) affecting functionality,
4. Patients with another disease (such as inflammatory diseases, polyneuropathy, brachial plexus lesion, loss of range of motion after trauma) affecting upper extremity functions.
5. Patients diagnosed with secondary Parkinson's disease
6. Patients with acute neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-04-25 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
improvement in hand functions | 3 months
  The Movement Disorder Society-Sponsored Revision of the Unified, which is used to evaluate the symptoms and signs of Parkinson's Disease, consists of a total of 4 chapters and 42 items. Each item is scored between 0 (normal) and 4 (most severe). The scores obtained are evaluated as a percentage. As the total score increases, it is understood that the mental status for the first part and the functional status for the other parts are worse. In this study, the motor part of the evaluation scale will be used. The patients will be evaluated three times. Once in the beginning (before the study), second evaluation will be made in the 1st month after the treatment and the 3rd month after the treatment the 3rd evaluation will be made. The change in the results of the scale (The Movement Disorder Society-Sponsored Revision of the Unified) evaluating the improvement in hand functions will be evaluated.

SECONDARY OUTCOMES:
Hand and Finger Grip Strength | 3 months
  Hand rough grip strength will be measured with a Jamar hydraulic hand dynamometer. A pinchmeter will be used for lateral, tip and triple grip measurement.
  The Jamar dynamometer has five stages. Measurements will be made in the position of the jamar suitable for the hand size of the patients, in the dominant extremity, with the patients in an upright position, shoulder adduction, elbow 90 degrees flexion, anterior colmidrotation and wrist 30 degrees extension, and maximum voluntary grasping will be requested from the patients. Measurements will be made 3 times and the average value will be recorded in kilograms. The patients will be evaluated three times. Once in the beginning (before the study), second evaluation will be made in the 1st month after the treatment and the 3rd month after the treatment the 3rd evaluation will be made. The change in the Hand and Finger Grip Strength will be evaluated.
quality of life | 3 months
  Parkinson's Disease questionnaire; It consists of eight sections and thirty-nine questions: mobility 10 questions, activities of daily living 6 questions, stigma 4 questions, emotional status 6 questions, cognition 4 questions, social support 3 questions, physical discomfort 3 questions, communication 3 questions. Each question is scored between 0 and 4. It is expressed as '0 never, 1 rarely, 2 sometimes, 3 often, 4 always'. The total value obtained is converted into points between 0-100. A low score indicates a good quality of life, and a high score indicates a poor quality of life.
  The patients will be evaluated three times. Once in the beginning (before the study), second evaluation will be made in the 1st month after the treatment and the 3rd month after the treatment the 3rd evaluation will be made. The change in the results of the scale (Parkinson's Disease questionnaire) evaluating the quality of life will be evaluated.
dexterity | 3 months
  Nine-hole peg test will be used for the evaluation of hand dexterity. Nine-hole peg test consists of nine small sticks and a board with nine holes on which these sticks can be placed. Patients will be asked to sit at the table and insert the sticks into the holes one by one as quickly as possible, and then collect them again. The elapsed time will be measured with recorded in seconds.
  The patients will be evaluated three times. Once in the beginning (before the study), second evaluation will be made in the 1st month after the treatment and the 3rd month after the treatment the 3rd evaluation will be made. The change in the hand dexterity will be evaluated.
dexterity | 3 months
  Minnesota Manual Dexterity test will be used for the evaluation of hand dexterity. The test consisted of 20 movable discs that could go from one hole to another. Removing, turning and placing the discs from the cavities was performed bilaterally in the right and left upper extremities, and the result was recorded in 'seconds'.
  The patients will be evaluated three times. Once in the beginning (before the study), second evaluation will be made in the 1st month after the treatment and the 3rd month after the treatment the 3rd evaluation will be made. The change in the hand dexterity will be evaluated.
dexterity | 3 months
  Box and block test will be used for the evaluation of hand dexterity. In the box and block test, there are 150 cubes in total in a box with a two-sided compartment. The cubes are 2.5 cm. edged. The patient is asked to move the cubes from one compartment to the other compartment one by one. The number of cubes carried in 60 seconds gives the test score.
  The patients will be evaluated three times. Once in the beginning (before the study), second evaluation will be made in the 1st month after the treatment and the 3rd month after the treatment the 3rd evaluation will be made. The change in the hand dexterity will be evaluated.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bonassi G, Pelosin E, Ogliastro C, Cerulli C, Abbruzzese G, Avanzino L. Mirror Visual Feedback to Improve Bradykinesia in Parkinson's Disease. Neural Plast. 2016;2016:8764238. doi: 10.1155/2016/8764238. Epub 2016 Aug 1. PMID 27563470
- [Background] Temporiti F, Adamo P, Cavalli E, Gatti R. Efficacy and Characteristics of the Stimuli of Action Observation Therapy in Subjects With Parkinson's Disease: A Systematic Review. Front Neurol. 2020 Aug 13;11:808. doi: 10.3389/fneur.2020.00808. eCollection 2020. PMID 32903559
- [Background] Carod-Artal FJ, Vargas AP, Martinez-Martin P. Determinants of quality of life in Brazilian patients with Parkinson's disease. Mov Disord. 2007 Jul 30;22(10):1408-1415. doi: 10.1002/mds.21408. PMID 17516479